CLINICAL TRIAL: NCT05523479
Title: The Maximizing Extubation Outcomes Through Educational and Organizational Research (METEOR) Trial
Acronym: METEOR
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Timothy Girard, MD, MSCI, Professor of Critical Care Medicine, University of Pittsburgh
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY20100469; U01HL159882 (NIH)
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Acute Respiratory Failure; Airway Extubation
Keywords: Interprofessional Education; Clinical Protocols; Noninvasive Ventilation; Oxygen Inhalation Therapy
MeSH Terms: interventions — Clinical Protocols; Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: The METEOR Trial is a batched stepped wedge cluster randomized type 2 hybrid implementation-effectiveness trial. ICUs are randomized rather than individuals, and each ICU will cross over from control to intervention at a randomized timepoint. The trial will employ three variations on the traditional stepped wedge design:
  1. A factorial design will be used to estimate the effects of two implementation strategies (IPE and a clinical protocol) separately as well as together.
  2. A concurrent design will be used to compare two post-extubation strategies (HFNC for all patients vs. NIV for high-risk patients and HFNC for low-risk patients) with conventional post-extubation oxygen therapy and with each other.
  3. A batched design allows for the recruitment of clusters (i.e., ICUs) throughout the duration of the trial rather than requiring that all clusters commence participation in the trial at the same time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- Online education about risk-stratified post-extubation NIV/HFNC (Active Comparator): During this period, ICU providers receive traditional online education that demonstrates the evidence supporting use of preventive post-extubation respiratory support (NIV or HFNC) over conventional post-extubation oxygen and supports the implementation of risk-stratified, preventive post-extubation NIV/HFNC.
  Interventions: Behavioral: Traditional online education; Other: Risk-stratified preventive post-extubation noninvasive ventilation (NIV) or high-flow nasal cannula oxygen (HFNC)
- Interprofessional education about risk-stratified post-extubation NIV/HFNC (Active Comparator): During this period, ICU providers receive interprofessional education that demonstrates the evidence supporting use of preventive post-extubation respiratory support (NIV or HFNC) over conventional post-extubation oxygen and supports the implementation of risk-stratified, preventive post-extubation NIV/HFNC.
  Interventions: Behavioral: Interprofessional education; Other: Risk-stratified preventive post-extubation noninvasive ventilation (NIV) or high-flow nasal cannula oxygen (HFNC)
- Clinical protocol about risk-stratified post-extubation NIV/HFNC (Active Comparator): During this period, ICU providers deploy a clinical protocol that supports the implementation of risk-stratified, preventive post-extubation NIV/HFNC.
  Interventions: Behavioral: Clinical protocol; Other: Risk-stratified preventive post-extubation noninvasive ventilation (NIV) or high-flow nasal cannula oxygen (HFNC)
- Interprofessional education plus clinical protocol about risk-stratified post-extubation NIV/HFNC (Active Comparator): During this period, ICU providers receive interprofessional education and use a clinical protocol that supports the implementation of risk-stratified, preventive post-extubation NIV/HFNC.
  Interventions: Behavioral: Interprofessional education; Behavioral: Clinical protocol; Other: Risk-stratified preventive post-extubation noninvasive ventilation (NIV) or high-flow nasal cannula oxygen (HFNC)
- Online education about post-extubation HFNC (Active Comparator): During this period, ICU providers receive traditional online education that demonstrates the evidence supporting use of preventive post-extubation respiratory support (NIV or HFNC) over conventional post-extubation oxygen and supports the implementation of preventive post-extubation HFNC for all eligible patients.
  Interventions: Behavioral: Traditional online education; Other: Preventive post-extubation high-flow nasal cannula oxygen (HFNC)
- Interprofessional education about post-extubation HFNC (Active Comparator): During this period, ICU providers receive interprofessional education that demonstrates the evidence supporting use of preventive post-extubation respiratory support (NIV or HFNC) over conventional post-extubation oxygen and supports the implementation of preventive post-extubation HFNC for all eligible patients.
  Interventions: Behavioral: Interprofessional education; Other: Preventive post-extubation high-flow nasal cannula oxygen (HFNC)
- Clinical protocol about post-extubation HFNC (Active Comparator): During this period, ICU providers deploy a clinical protocol that supports the implementation of preventive post-extubation HFNC for all eligible patients.
  Interventions: Behavioral: Clinical protocol; Other: Preventive post-extubation high-flow nasal cannula oxygen (HFNC)
- Interprofessional education plus clinical protocol about post-extubation HFNC (Active Comparator): During this period, ICU providers receive interprofessional education and use a clinical protocol that supports the implementation of preventive post-extubation HFNC for all eligible patients.
  Interventions: Behavioral: Interprofessional education; Behavioral: Clinical protocol; Other: Preventive post-extubation high-flow nasal cannula oxygen (HFNC)
- Usual care (No Intervention): During this period, ICU providers receive no structured education about preventive, post-extubation respiratory support therapies

INTERVENTIONS:
Behavioral: Traditional online education — A 30-60 minute, online, interactive, educational video that is customized to each provider type and offered with provider-specific continuing education credits
  Arms: Online education about post-extubation HFNC; Online education about risk-stratified post-extubation NIV/HFNC
Behavioral: Interprofessional education — Interprofessional education (IPE) consists of both classroom-based IPE and just-in-time IPE. In classroom-based IPE, a trained physician educator with content expertise who works in the ICU leads a 60-to-90-minute, in-person, IPE workshop consisting of a 30-minute didactic session and a 30-to-60-minute small group session, during which participants work together to apply the content to authentic cases. The workshops, which are designed according to modern principles of adult learning and IPE, present the rationale and evidence supporting the preventive, post-extubation therapies. They are specifically designed to foster authenticity, reinforce role identity, and relate the content to life experience. In just-in-time IPE, trained local champions meet with the interprofessional ICU team each morning to identify eligible patients and, as needed, briefly review the evidence supporting proper use of the assigned preventive, post-extubation strategy.
  Arms: Interprofessional education about post-extubation HFNC; Interprofessional education about risk-stratified post-extubation NIV/HFNC; Interprofessional education plus clinical protocol about post-extubation HFNC; Interprofessional education plus clinical protocol about risk-stratified post-extubation NIV/HFNC
Behavioral: Clinical protocol — An "adequately explicit" protocol provides specific rules for use of the preventive, post-extubation therapy based on patient data. A "ready-to-customize" version of the protocol with instructions to work with key local stakeholders to revise the protocol, accounting for local needs and resources, is provided. After local customization, a local champion then disseminates the protocol based on local practices.
  Arms: Clinical protocol about post-extubation HFNC; Clinical protocol about risk-stratified post-extubation NIV/HFNC; Interprofessional education plus clinical protocol about post-extubation HFNC; Interprofessional education plus clinical protocol about risk-stratified post-extubation NIV/HFNC
Other: Risk-stratified preventive post-extubation noninvasive ventilation (NIV) or high-flow nasal cannula oxygen (HFNC) — Preventive post-extubation NIV for high-risk patients and preventive post-extubation HFNC for low-risk patients
  Arms: Clinical protocol about risk-stratified post-extubation NIV/HFNC; Interprofessional education about risk-stratified post-extubation NIV/HFNC; Interprofessional education plus clinical protocol about risk-stratified post-extubation NIV/HFNC; Online education about risk-stratified post-extubation NIV/HFNC
Other: Preventive post-extubation high-flow nasal cannula oxygen (HFNC) — Preventive post-extubation HFNC for all eligible patients (without risk stratification)
  Arms: Clinical protocol about post-extubation HFNC; Interprofessional education about post-extubation HFNC; Interprofessional education plus clinical protocol about post-extubation HFNC; Online education about post-extubation HFNC

SUMMARY:
The METEOR Trial will compare four implementation strategies-traditional online education, protocol-directed care, interprofessional education, and a combination of protocol-directed care and interprofessional education-to test the hypotheses that interprofessional education is superior to traditional online education as an implementation strategy in the intensive care unit (ICU) and the benefits of interprofessional education are increased when interprofessional education is paired with a clinical protocol. Additionally, the trial will also test the hypothesis that preventive post-extubation NIV for high-risk patients and preventive post-extubation HFNC for low-risk patients are both superior to current clinical practice (i.e., conventional post-extubation oxygen therapy).

DETAILED DESCRIPTION:
Nearly one million patients require invasive mechanical ventilation for acute respiratory failure in the United States each year. Most of these patients will recover to the point of extubation, yet even those who are extubated remain vulnerable to complications and poor outcomes. Multiple high-profile randomized controlled trials have shown that two preventive post-extubation respiratory therapies-noninvasive ventilation (NIV) and high-flow nasal cannula oxygen (HFNC)-can prevent recurrent respiratory failure, reintubation, and death in this population. Despite this evidence, however, these therapies remain severely underutilized, leading to preventable morbidity and mortality. To address this implementation gap, the investigators will conduct the Maximizing Extubation outcomes Through Educational and Organizational Research (METEOR) Trial, a cluster-randomized, stepped-wedge, type 2 hybrid effectiveness-implementation trial of interprofessional education about preventive post-extubation NIV and HFNC with and without clinical protocols. The METEOR Trial was designed based on extensive preliminary studies, during which the investigators identified barriers to adoption of preventive post-extubation respiratory care and pilot tested interprofessional education as an implementation strategy in the ICU. These studies revealed that a major barrier to implementation is the lack of a shared understanding about the value of these therapies within the interprofessional ICU team; a theory-based interprofessional education intervention designed to create a shared understanding and support "transactive memory" among team members is both feasible and acceptable; and interprofessional education can be strengthened by linking it with a clinical protocol. During the METEOR Trial, the investigators will randomize ICUs to one of four implementation strategies: an active control, protocol-directed care, interprofessional education, or a combination of protocol-directed care and interprofessional education. In parallel, the investigators will randomize ICUs to one of two clinical strategies, one emphasizing either post- extubation NIV or HFNC based on patient risk vs. one emphasizing post-extubation HFNC for all patients.

ELIGIBILITY:
Inclusion Criteria:

* All adults treated with invasive mechanical ventilation >24 hours in participating ICUs

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13018 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Rate of use of post-extubation NIV or HFNC among eligible participants (primary implementation outcome) | 60 days after initiating invasive mechanical ventilation
  Defined the number of participants who received post-extubation NIV or HFNC divided by the number of participants eligible for post-extubation NIV or HFNC
In-hospital mortality truncated at 60 days from intubation (primary clinical outcome) | 60 days after initiating invasive mechanical ventilation
  Defined as the number of participants who died during hospitalization

SECONDARY OUTCOMES:
Number of eligible participants receiving care from providers who completed an implementation intervention | Up to 3 years
  Defined as the total number of participants who received care from ICU providers (physicians, nurses, and/or respiratory therapists) who completed an implementation intervention (traditional online education, interprofessional education, and/or clinical protocol)
Use of post-extubation NIV or HFNC among eligible participants 6 months after the implementation intervention (IPE plus protocol) is fully deployed | 6 months after the implementation intervention (IPE plus protocol) is fully deployed
  Defined the number of participants who received post-extubation NIV or HFNC divided by the number of participants eligible for post-extubation NIV or HFNC during the one-month period beginning 6 months after the implementation intervention (IPE plus protocol) is fully deployed
90-day survival | 90 days after initiating invasive mechanical ventilation
  Defined as time from initiating invasive mechanical ventilation to the date of death from any cause or last known follow-up (censored)
ICU length of stay | 60 days after initiating invasive mechanical ventilation
  Defined as time from the time of initiating invasive mechanical ventilation to successful discharge from the ICU, where "successful" indicates that discharge was followed by at least 48 hours alive without ICU readmission
Hospital length of stay | 60 days after initiating invasive mechanical ventilation
  Defined as time from the time of initiating invasive mechanical ventilation to successful hospital discharge, where "successful" indicates that discharge was followed by at least 48 hours alive without hospital readmission
Post-extubation respiratory failure | 60 days after initiating invasive mechanical ventilation
  Defined as reintubation and resumption of invasive mechanical ventilation during the 48 hours after extubation
Duration of mechanical ventilation | 60 days after initiating invasive mechanical ventilation
  Defined as time from the time of initiating invasive mechanical ventilation to successful extubation, where "successful" indicates that extubation was followed by at least 48 hours alive without reintubation
28-day ventilator-free days (VFDs) | 28 days after initiating invasive mechanical ventilation
  Defined as the number of days a participant was breathing without assistance from the day they of intubation (initiating invasive mechanical ventilation) to 28 days later, where "breathing without assistance" indicates that discontinuation of assisted breathing was followed by at least 48 hours alive without reintubation
Ventilator-associated events (VAEs) | Up to 60 days after initiating invasive mechanical ventilation
  Defined as the number of participants who have a VAE according to Centers of Disease Control and Prevention (CDC) criteria divided by the number of participants who received invasive mechanical ventilation
Organ failure (daily SOFA) | Up to 60 days after initiating invasive mechanical ventilation
  Defined as mean daily sequential organ failure assessment (SOFA) score from initiating invasive mechanical ventilation to up to 60 days later

CONTACTS AND LOCATIONS:
Overall Officials: Timothy D Girard, MD, MSCI, Principal Investigator — University of Pittsburgh
Locations (15):
- United States (15):
  - UPMC Carlisle, Carlisle, Pennsylvania
  - UPMC Hanover, Hanover, Pennsylvania
  - UPMC Harrisburg, Harrisburg, Pennsylvania
  - UPMC Community Osteopathic, Harrisburg, Pennsylvania
  - UPMC West Shore, Mechanicsburg, Pennsylvania
  - UPMC East, Monroeville, Pennsylvania
  - UPMC Jameson, New Castle, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - UPMC Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - UPMC St. Margaret, Pittsburgh, Pennsylvania
  - UPMC Mercy, Pittsburgh, Pennsylvania
  - UPMC Shadyside, Pittsburgh, Pennsylvania
  - UPMC Passavant, Pittsburgh, Pennsylvania
  - UPMC Memorial, York, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The University of Pittsburgh will comply with applicable NIH guidelines on data sharing as published online. The investigators will make scientific data as widely and freely available as possible while safeguarding the privacy of participants and protecting confidential and proprietary data. Data will be shared as elements that meet or exceed the HIPAA Privacy Rule definition of "safe harbor de-identified" data, so that the rights and privacy of human subjects who participate in research are protected at all times. Principles and guidelines as outlined by the NIH Office of Technology Transfer will be observed in sharing all scientific resources.
Supporting Information: Study Protocol, SAP
Time Frame: Deidentified individual participant data will be made available to investigators who provide a methodologically sound proposal to achieve the aims of the approved proposal. Data will be available as soon as possible but no later than within one year of the completion of the funded project period or upon acceptance of the data for publication, whichever is earlier.
Access Criteria: Proposals should be directed to Timothy Girard at timothy.girard@pitt.edu. To gain access, data requestors will need to sign a data use agreement.

REFERENCES:
- [Background] Ouellette DR, Patel S, Girard TD, Morris PE, Schmidt GA, Truwit JD, Alhazzani W, Burns SM, Epstein SK, Esteban A, Fan E, Ferrer M, Fraser GL, Gong MN, Hough CL, Mehta S, Nanchal R, Pawlik AJ, Schweickert WD, Sessler CN, Strom T, Kress JP. Liberation From Mechanical Ventilation in Critically Ill Adults: An Official American College of Chest Physicians/American Thoracic Society Clinical Practice Guideline: Inspiratory Pressure Augmentation During Spontaneous Breathing Trials, Protocols Minimizing Sedation, and Noninvasive Ventilation Immediately After Extubation. Chest. 2017 Jan;151(1):166-180. doi: 10.1016/j.chest.2016.10.036. Epub 2016 Nov 3. PMID 27818331
- [Background] Rochwerg B, Brochard L, Elliott MW, Hess D, Hill NS, Nava S, Navalesi P Members Of The Steering Committee, Antonelli M, Brozek J, Conti G, Ferrer M, Guntupalli K, Jaber S, Keenan S, Mancebo J, Mehta S, Raoof S Members Of The Task Force. Official ERS/ATS clinical practice guidelines: noninvasive ventilation for acute respiratory failure. Eur Respir J. 2017 Aug 31;50(2):1602426. doi: 10.1183/13993003.02426-2016. Print 2017 Aug. PMID 28860265
- [Background] Granton D, Chaudhuri D, Wang D, Einav S, Helviz Y, Mauri T, Mancebo J, Frat JP, Jog S, Hernandez G, Maggiore SM, Hodgson CL, Jaber S, Brochard L, Trivedi V, Ricard JD, Goligher EC, Burns KEA, Rochwerg B. High-Flow Nasal Cannula Compared With Conventional Oxygen Therapy or Noninvasive Ventilation Immediately Postextubation: A Systematic Review and Meta-Analysis. Crit Care Med. 2020 Nov;48(11):e1129-e1136. doi: 10.1097/CCM.0000000000004576. PMID 32947472
- [Background] Sang L, Nong L, Zheng Y, Xu Y, Chen S, Zhang Y, Huang Y, Liu X, Li Y. Effect of high-flow nasal cannula versus conventional oxygen therapy and non-invasive ventilation for preventing reintubation: a Bayesian network meta-analysis and systematic review. J Thorac Dis. 2020 Jul;12(7):3725-3736. doi: 10.21037/jtd-20-1050. PMID 32802452
- [Background] Fernando SM, Tran A, Sadeghirad B, Burns KEA, Fan E, Brodie D, Munshi L, Goligher EC, Cook DJ, Fowler RA, Herridge MS, Cardinal P, Jaber S, Moller MH, Thille AW, Ferguson ND, Slutsky AS, Brochard LJ, Seely AJE, Rochwerg B. Noninvasive respiratory support following extubation in critically ill adults: a systematic review and network meta-analysis. Intensive Care Med. 2022 Feb;48(2):137-147. doi: 10.1007/s00134-021-06581-1. Epub 2021 Nov 25. PMID 34825256
- [Background] Argote L, Miron-Spektor E. Organizational learning: From experience to knowledge. Organization Science 2011;22:1123-37.
- [Background] Kasza J, Bowden R, Hooper R, Forbes AB. The batched stepped wedge design: A design robust to delays in cluster recruitment. Stat Med. 2022 Aug 15;41(18):3627-3641. doi: 10.1002/sim.9438. Epub 2022 May 21. PMID 35596691
- [Derived] Prendergast NT, Kahn JM, Angus DC, Argote L, Barnes B, Chang CH, Graff S, Hess DR, Onyemekwu CA, Rak KJ, Russell JL, Seaman JB, Toth KM, Girard TD. Maximizing Extubation Outcomes Through Educational and Organizational Research (METEOR) Trial: protocol for a batched, stepped-wedge, cluster-randomised, type 2 hybrid effectiveness-implementation trial. BMJ Open. 2025 Oct 23;15(10):e108956. doi: 10.1136/bmjopen-2025-108956. PMID 41130691